CLINICAL TRIAL: NCT03008681
Title: Oral Health-Related Quality of Life in Patients With Juvenile Idiopathic Arthritis and Temporomandibular Joint Disorders Evaluation After Treatment With a Functional Appliance
Brief Title: OHRQoL Evaluation After Functional Therapy in JIA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, DDS. PhD, University of Messina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-918
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Andresen functional removable orthodontic appliance (Experimental): All the enrolled patients was applied the Andresen Activator (a removable orthodontic appliance) 12-14 hours in a day in total.
  Functional appliances helped the movement of the teeth, with the achievement of good facial muscle function. All patients in the cohort were treated with the andresen actovator appliancev for deep bite and class II malocclusion correction.
  The appliances were individually manufactured of acrylic resin, with a central screw and a vestibular arch, fabricated through a wax bite registration; the patient was guided to close the mouth in mandibular protrusion with coincidence of the upper and lower midlines. The registration bite was very thin in order to obtain a minimum vertical dimension. The activator was modified every three months increasing its posterior vertical dimension in order to stimulate the mandibular ramus growth thanks to the dislocation of the mandibular condyle.
  Interventions: Device: Andresen functional removable orthodontic appliance

INTERVENTIONS:
Device: Andresen functional removable orthodontic appliance — Included patients were treated for 24 months with a Functional removable orthodontic appliance, the Andresen activator. The initial checks were performed after 6 weeks with subsequent checks being carried out every 8th week, with the final follow-up at 24 months. The patient underwent functional treatment using the activator described in the protocol with midlines coincidence.
  Other Names: Andresen Activator

SUMMARY:
The aim of the study was to determine the changes in Oral Health-Related Quality of Life (OHRQoL) in patients with juvenile idiopathic arthritis (JIA) and temporomandibular joint (TMJ) disorders who underwent functional therapy for 24 months to assess the age and sex group in which the functional therapy was most effective.

DETAILED DESCRIPTION:
This prospective interventional study included 93 patients with JIA and TMJ disorders at the start of functional orthodontic therapy. Children were prospectively followed in the 24 months of treatment and completed the Oral Health Impact Profile (OHIP-14) before treatment (T0), and at 6 months (T1), 12 months (T2), and 24 months (T3) after the start of therapy.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were:

* JIA with unilateral or bilateral TMJ arthritis treated with a functional appliance;
* Clear signs or symptoms of TMJ arthritis based on clinical and radiological examination.
* No administration of intra-articular TMJ steroid injections throughout the course of the orthopaedic functional treatment.

Exclusion Criteria:

* previous orthodontic treatment;
* history of maxillofacial surgery;
* genetic diseases, syndromes, other congenital deformities or any concurrent medical condition.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2004-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
TMJ disorder cessation | 24 months
  TMJ disorder and clinical mandibular symmetry was achieved or if mandibular growth was estimated as ceased.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, DDS, Study Director — University of Messina
Locations (1):
- University of Messina, Messina, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isola G, Perillo L, Migliorati M, Matarese M, Dalessandri D, Grassia V, Alibrandi A, Matarese G. The impact of temporomandibular joint arthritis on functional disability and global health in patients with juvenile idiopathic arthritis. Eur J Orthod. 2019 Mar 29;41(2):117-124. doi: 10.1093/ejo/cjy034. PMID 29878100